CLINICAL TRIAL: NCT06188156
Title: Analgesic Efficacy of Ultrasound Guided Serratus Anterior Plane Block and Pectoral Nerve Block II Compared to Thoracic Epidural Block After Unilateral Modified Radical Mastectomy
Brief Title: Analgesic Efficacy of Ultrasound Guided Serratus Anterior Plane Block and Pectoral Nerve Block II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, mohamed A Aboelsuod, MD, Assistant Professor of Anesthesia, intensive care and pain management Faculty of Medicine, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ahmed Elbasuni Ali
Record Dates: First submitted 2023-12-10; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Anesthesia; Radical Mastectomy
Keywords: thoracic epidural blockage; Ultrasound Guided Serratus Anterior Plane Block; Pectoral Nerve Block II; Radical Mastectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Thoracic Epidural Block(Group 1) (Active Comparator): About 33 Patients will receive thoracic epidural block with an injection of a single shot of 15ml of 0.25% bupivacaine between T4 and T5 vertebrae.
  Interventions: Procedure: Anethesia
- Ultrasound Guided Sserratus Anterior Plane Block (Group 2) (Active Comparator): About 33 Patients will receive Ultrasound Guided Sserratus Anterior Plane Block( SAPB) with an injection of 30 ml bupivacaine 0.25% .
  Interventions: Procedure: Anethesia
- Ultrasound Guided Pectoral Nerve Block (Group 3) (Active Comparator): About 33 Patients will receive Ultrasound Guided Pectoral Nerve Block ( PECS II) with an injection of 20 ml bupivacaine 0.25% of pectoral-minor above the Serratus anterior muscle.
  Interventions: Procedure: Anethesia

INTERVENTIONS:
Procedure: Anethesia — To assess the effectiveness of thoracic epidural blockage versus ultrasonic guided PECS II block versus ultrasound guided serratus anterior plane block for postoperative pain management in modified radical mastectomy.

SUMMARY:
Modified Radical Mastectomy accounts for 31% of all breast surgeries and considered the fundamental surgical management for breast cancer. Nearly 40-60% of patients experience severe acute postoperative pain. This pain might persist for 6-12 months and result in post-mastectomy pain syndrome and complex regional pain syndrome (causalgia)

DETAILED DESCRIPTION:
There are some local or regional nerve blocks in breast surgeries performed as core components of multimodal analgesia and enhanced recovery after surgery (ERAS), including thoracic epidural (TEB), interscalene brachial plexus, paravertebral, ultrasound-guided pectoral nerve block ( PECS II ), ultrasound-guided serratus anterior plane block (SAPB) and erector spinae plane block .

Thoracic epidural (TEB) is the gold standard technique following breast surgery, but there is still a problem with the adequacy of thoracic and axillary blockage during lymph node dissection .

Modified PECS's block" or PECS block type II aimed to block the axilla that is vital for axillary clearances and the intercostal nerves, necessary for wide excisions which can provide analgesia after breast surgery.

In the ultrasound-guided serratus anterior plane block (SAPB), the local anesthetic (LA) is injected in the compartment between the serratus anterior and latissimus dorsi muscles. SAPB anesthetizes the intercostobrachial nerve, lateral cutaneous branches of the intercostal nerves (T3-T9), long thoracic nerve, and thoracodorsal nerve thus providing analgesia for breast and lateral thoracic wall surgeries

ELIGIBILITY:
Inclusion Criteria:

* Women aged 35-65 years.
* BMI 18.5 - 25 kg/m2.
* American Society of Anesthesiologists (ASA) I-II.

Exclusion Criteria:

* Patient refusal.
* Coagulopathy.
* Mental and psychiatric disorders.
* History of chronic pain.
* Hypersensitivity or contraindication to any of study drugs
* Previous chemotherapy.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Measurement of Post-operative Pain | First 24-hour analgesic after Mastectomy
  Assessment of the pain post-operatively in patients with pain assessed by VAS score : Total scores vary from 0 to 10 in this method, with a higher score indicating more severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Aldine Mahmoud Said, Professor, Study Chair — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No